CLINICAL TRIAL: NCT00731393
Title: To Determine the Immunogenicity and Reactogenicity of a Thiomersal Free Trivalent Influenza Split Vaccine 2003/2004 or of GSK Biologicals' Standard Formulation Influsplit SSW®/Fluarix™ 2003/2004 in Children Aged From 6 Months Until 6 Years
Brief Title: Immuno & Reacto of TF Trivalent Influenza Split Vaccine 2003/04 or of Std Formulation Influsplit SSW®/Fluarix™ 2003/04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 100351
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Influenza
Keywords: Thiomersal-free influenza split vaccine 2003/2004; Influsplit SSW®/Fluarix™ 2003/2004; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Subjects aged between 6 months and 3 years.
  Interventions: Biological: Thiomersal free trivalent influenza split vaccine 2003/2004
- Group B (Experimental): Subjects aged 3 to 6 years.
  Interventions: Biological: Thiomersal free trivalent influenza split vaccine 2003/2004
- Group C (Active Comparator): Subjects aged between 6 months and 3 years.
  Interventions: Biological: GlaxoSmithKline Biologicals' Influsplit SSW®/Fluarix™ 2003/2004
- Group D (Active Comparator): Subjects aged 3 to 6 years.
  Interventions: Biological: GlaxoSmithKline Biologicals' Influsplit SSW®/Fluarix™ 2003/2004

INTERVENTIONS:
Biological: Thiomersal free trivalent influenza split vaccine 2003/2004 — 2 doses, intramuscular injection
  Arms: Group A; Group B
Biological: GlaxoSmithKline Biologicals' Influsplit SSW®/Fluarix™ 2003/2004 — 2 doses, intramuscular injection
  Other Names: Thiomersal free trivalent influenza split vaccine 2003/2004
  Arms: Group C; Group D

SUMMARY:
The aim of the present study is to assess the reactogenicity and immunogenicity of a thiomersal-free influenza vaccine. For comparison, a group of subjects is administered the standard formulation of Influsplit SSW® 2003/2004.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose parents/guardians the investigator believes can and will comply with the requirements of the protocol
* Male or female children over 6 months of age at the time of vaccination, but who are not yet 6 years old.
* All children included in the study must never have been given a prophylactic influenza inoculation.
* Written consent to vaccination must be available from both parents or only the single parent after the parents/guardians have been briefed on the study in an understandable language.

Exclusion Criteria:

* Use of study or unlicensed medication or administration of a vaccine other than the study vaccine within 30 days preceding vaccination and/or during the study period until 30 days after administration of the second vaccine dose.
* Acute disease at the beginning of the study
* Acute clinically significant changes in the lungs, cardiovascular system, liver or kidney function, identified by physical examination or laboratory tests.
* Known allergic reactions that might have been caused by one or more components of the vaccine.
* Administration of immunoglobulins and/or other blood products within 3 months before the beginning of the study or planned administration during the study period.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2003-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
GMT of the haemagglutination-inhibiting (HI) antibodies and calculation of seroconversion factor, seroconversion rate & seroprotection rate, checked against CHMP criteria (for 18 - 60 years old); seroprotection power is also calculated. | On Day 21 (+- 2) after the second vaccination

SECONDARY OUTCOMES:
Descriptive comparison of the occurrence and severity of solicited local and general symptoms | Within 4 days after each vaccination
Descriptive comparison of the occurrence, severity and relationship to vaccination of unsolicited signs and symptoms | Within 30 days after each vaccination
Descriptive comparison of the occurrence, severity and relationship to vaccination of serious adverse events (SAEs). | Throughout the study
GMT of the HI antibodies in each case against the 3 influenza virus strains of the vaccine separately for both age groups. | On Day 21 (+- 2), Month 3 and Month 6 after the second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Germany (10):
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bischofswerda, Saxony
  - GSK Investigational Site, Coswig, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100351 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register